CLINICAL TRIAL: NCT02241889
Title: A Randomized, Three-way, Cross-over Study to Assess the Efficacy of a Bi-hormonal Closed-loop System With vs Without Exercise Announcement vs Open-loop Therapy in Reducing Exercise-related Hypoglycemia
Brief Title: Three-way, Cross-over Closed-loop Exercise Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Jessica Castle, Assistant Professor, Oregon Health and Science University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: DP3-2014
Record Dates: First submitted 2014-09-12; First posted 2014-09-16 (Estimated); Results first posted 2017-05-22 (Actual); Last update posted 2017-05-22 (Actual); Status verified 2017-04

CONDITIONS: Type 1 Diabetes
Keywords: diabetes; closed-loop; bi-hormonal; exercise
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Standard Insulin Pump Therapy (Active Comparator): Subjects will undergo 21 hour study with exercise using Insulin pump therapy and managing their blood glucose as they normally would.
  Interventions: Device: Insulin pump therapy
- Closed-loop without adjustment (Experimental): Subjects will undergo 21 study using the Closed-loop Artificial Pancreas Controller to manage blood sugar. Exercise will not be annouced to the controller and no adjustments to insulin and glucagon delivery will be made.
  Interventions: Device: Closed-loop Artificial Pancreas Controller
- Closed-loop with adjustment (Experimental): Subjects will undergo 21 hour study using the Closed-loop Artificial Pancreas Controller to manage blood sugar. Exercise will be annouced to the controller and adjustments to insulin and glucagon delivery will be made.
  Interventions: Device: Closed-loop Artificial Pancreas Controller

INTERVENTIONS:
Device: Insulin pump therapy — Subject's own insulin pump will be used to manage blood glucose.
  Arms: Standard Insulin Pump Therapy
Device: Closed-loop Artificial Pancreas Controller — Closed-loop Artificial Pancreas Controller includes insulin and glucagon delivery algorithm implemented on a smart phone, utilizing sensor glucose values from a Dexcom G4 sensor and sending delivery commands to two Tandem t:slim insulin pumps, one filled with insulin and one with glucagon.
  Arms: Closed-loop with adjustment; Closed-loop without adjustment

SUMMARY:
Blood glucose control systems that utilize both insulin and glucagon to manage blood sugar are paving the way to revolutionize the management of this disease. The benefit of improved control of blood sugar levels compared to standard insulin pump therapy has already been demonstrated. However, the risk of low blood sugar in type 1 diabetes increases considerably during exercise. The investigators research group has shown that small doses of glucagon can prevent low blood sugar when used in a blood sugar control system in patients with type 1 diabetes. However, as insulin sensitivity changes occur very rapidly during exercise, the ability to recognize the onset of physical activity in order to appropriately adjust the insulin and glucagon delivery is vital to helping prevent exercise-induced hypoglycemia.

The purpose of this study is to test how well a new modified blood sugar control system controls blood sugar during exercise compared to: 1) the current system without modifications and 2) standard insulin pump therapy.

DETAILED DESCRIPTION:
Subjects will exercise during three study visits. During one visit, blood sugar will be controlled using standard insulin pump therapy. The investigators blood glucose control system will manage blood sugar for subjects during the other visits, with exercise announcement with insulin and glucagon delivery modifications during one visit. Treatment order will be randomized. Heart rate and accelerometry data will also be collected during each visit for the purposes of designing an exercise detection system for future studies.

Each subject will be asked to undergo an eligibility screening and to sign a consent form before any study procedures take place. At the screening appointment, after the consent form is signed, blood will be drawn for laboratory tests and a brief physical exam will be performed. An EKG and VO2max test will be completed at screening. Subjects that are enrolled in the study will come in for a sensor insertion visit up to 72 hours before each study visit. Subjects will undergo three 21-hour studies at an OHSU clinic or the OHSU clinical research center. Subjects will arrive at the research center at 8pm. Approximately 2 hours after a low-carbohydrate breakfast on Day 2, subjects will exercise for 45 minutes at 60% of their VO2max determined at screening. Three hours after completion of exercise, subjects will eat lunch. The study will end ~5 hours after lunch. Capillary blood glucose (CBG) will be measured every 2 hours during the day, every 3 hours at night and before and after exercise for studies using the blood glucose control system with subjects blinded to the CBG values. For studies using insulin pump therapy, the subject will sample CBG four times during the day as well as before and after exercise. Study staff will monitor studies remotely using a cloud server. An investigator or nurse practitioner with a specialty in endocrinology or internal medicine will be on site (located within the same complex) at all times.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of type 1 diabetes mellitus for at least 1 year.
* Male or female subjects 21 to 45 years of age.
* Physically willing and able to perform 45 min of exercise (as determined by the investigator after reviewing the subjects activity level)
* Current use of an insulin pump.
* Willingness to follow all study procedures, including attending all clinic visits.
* Willingness to sign informed consent and HIPAA documents.

Exclusion Criteria:

* Female of childbearing potential who is pregnant or intending to become pregnant or breast-feeding, or is not using adequate contraceptive methods. Acceptable contraception includes birth control pill / patch / vaginal ring, Depo-Provera, Norplant, an IUD, the double barrier method (the woman uses a diaphragm and spermicide and the man uses a condom), or abstinence.
* Any cardiovascular disease, defined as a clinically significant EKG abnormality at the time of screening or any history of: stroke, heart failure, myocardial infarction, angina pectoris, or coronary arterial bypass graft or angioplasty. Diagnosis of 2nd or 3rd degree heart block or any non-physiological arrhythmia judged by the investigator to be exclusionary.
* Renal insufficiency (GFR < 60 ml/min, using the MDRD equation as report by the OHSU laboratory).
* Impaired liver function, defined as AST or ALT ≥2.5 times upper limit of normal, according to OHSU laboratory reference ranges.
* Hematocrit of less than or equal to 34%.
* History of severe hypoglycemia during the past 12 months prior to screening visit or hypoglycemia unawareness as judged by the investigator.
* Adrenal insufficiency.
* Any active infection.
* Known or suspected abuse of alcohol, narcotics, or illicit drugs.
* Seizure disorder.
* Active foot ulceration.
* Severe peripheral arterial disease characterized by ischemic rest pain or severe claudication.
* Major surgical operation within 30 days prior to screening.
* Use of an investigational drug within 30 days prior to screening.
* Chronic usage of any immunosuppressive medication (such as cyclosporine, azathioprine, sirolimus, or tacrolimus).
* Bleeding disorder, treatment with warfarin, or platelet count below 50,000.
* Allergy to aspart insulin.
* Allergy to glucagon.
* Insulin resistance requiring more than 200 units per day.
* Need for uninterrupted treatment of acetaminophen.
* Current administration of oral or parenteral corticosteroids.
* Any life threatening disease, including malignant neoplasms and medical history of malignant neoplasms within the past 5 years prior to screening (except basal and squamous cell skin cancer).
* C peptide level of ≥0.5 ng/ml
* Any concurrent illness, other than diabetes, that is not controlled by a stable therapeutic regimen.
* Beta blockers or non-dihydropyridine calcium channel blockers.
* A positive response to any of the questions from the Physical Activity Readiness Questionnaire.
* Any clinically significant disease or disorder which in the opinion of the Investigator may jeopardize the subject's safety or compliance with the protocol.

Ages: 21 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2015-01; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Castle, MD, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health and Science University, Portland, Oregon, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- SAP, APN, APX (21 Hours): The randomization order for subjects in this arm was open loop (Sensor Augmented Pump SAP), closed loop (APN) and closed loop with exercise announcement (APX). Each visit was 21 hours.
- SAP, APX, APN (21 Hours): The randomization order for subjects in this arm was open loop (Sensor Augmented Pump SAP), closed loop with exercise announcement (APX), and closed loop (APN). Each visit was 21 hours.
- APN, SAP and APX (21 Hours): The randomization order for subjects in this arm was closed loop (APN), open loop (Sensor Augmented Pump SAP), and closed loop with exercise announcement (APX). Each visit was 21 hours.
- APN, APX, SAP (21 Hours): The randomization order for subjects in this arm was closed loop (APN), closed loop with exercise announcement (APX), and open loop (Sensor Augmented Pump SAP). Each visit was 21 hours.
- APX, SAP, APN (21 Hours): The randomization order for subjects in this arm was closed loop with exercise announcement (APX), open loop (Sensor Augmented Pump SAP) and closed loop (APN). Each visit was 21 hours.
- APX, APN, SAP (21 Hours): The randomization order for subjects in this arm was closed loop with exercise announcement (APX), closed loop (APN) and open loop (Sensor Augmented Pump SAP). Each visit was 21 hours.
Period: Overall Study
Arm/Group | SAP, APN, APX (21 Hours) | SAP, APX, APN (21 Hours) | APN, SAP and APX (21 Hours) | APN, APX, SAP (21 Hours) | APX, SAP, APN (21 Hours) | APX, APN, SAP (21 Hours)
Started | 4 | 4 | 3 | 3 | 5 | 4
Completed | 4 | 4 | 2 | 3 | 5 | 3
Not Completed | 0 | 0 | 1 | 0 | 0 | 1
Not completed — device issues | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Type 1 diabetics using an insulin pump
Groups:
- All Study Participants: All study participants underwent three 21 hour study visits using either standard of care insulin pump therapy, closed loop control, or closed loop control with adjustments to insulin and glucagon after exercise announcement. Treatment order was randomized.
Arm/Group | All Study Participants
Number analyzed (Participants) | 23
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 23
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 32 (7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 9
Region of Enrollment [Number; unit: participants]
  United States | 23

OUTCOME MEASURES:

1. Primary Outcome: Percent of Time With Sensed Glucose < 70 mg/dl
Description: Assess the percent of time that the Dexcom G4 or G4 Share reported sensor glucose values less than 70 mg/dl using Dexcom sensor downloads.
Time Frame: from start of exercise (~hour 12) until study completion (hour 21)
Population: Data was analyzed from 21 subjects that completed all 3 visits and visits went to completion. No data was analyzed from the two subjects that did not complete all visits.
Measure: Mean (95% Confidence Interval); unit: percentage of time
Groups:
- Closed-loop Without Adjustment: Subjects will undergo 21 hour study using the Closed-loop Artificial Pancreas Controller to manage blood sugar. Exercise will not be annouced to the controller and no adjustments to insulin and glucagon delivery will be made.
  Closed-loop Artificial Pancreas Controller: Closed-loop Artificial Pancreas Controller includes insulin and glucagon delivery algorithm implemented on a smart phone, utilizing sensor glucose values from a Dexcom G4 sensor and sending delivery commands to two Tandem t:slim insulin pumps, one filled with insulin and one with glucagon.
Arm/Group | Standard Insulin Pump Therapy | Closed-loop Without Adjustment | Closed-loop With Adjustment
Number analyzed (Participants) | 21 | 21 | 21
percentage of time | 0.9 [0.2 to 1.6] | 3.2 [0.9 to 5.5] | 0.3 [0.0 to 0.8]

2. Primary Outcome: Percent of Time With Sensed Glucose Between 70-180 mg/dl
Description: Assess the percent of time that the Dexcom G4 or G4 Share reported sensor glucose values between 70-180 mg/dl using Dexcom sensor downloads.
Time Frame: from start of exercise (~hour 12) until study completion (hour 21)
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: percent of time
Arm/Group | Standard Insulin Pump Therapy | Closed-loop Without Adjustment | Closed-loop With Adjustment
Number analyzed (Participants) | 21 | 21 | 21
percent of time | 67.6 [59.5 to 75.7] | 72.5 [66.3 to 78.8] | 67.3 [60.2 to 74.5]

3. Secondary Outcome: Mean of the Mean Sensed Glucose Per Participant
Description: Assess the mean sensed glucose per participant using Dexcom sensor downloads.
Time Frame: Entire 21 hour study duration excluding the first four hours
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: mg/dl
Arm/Group | Standard Insulin Pump Therapy | Closed-loop Without Adjustment | Closed-loop With Adjustment
Number analyzed (Participants) | 21 | 21 | 21
mg/dl | 8.6 [7.9 to 9.2] | 8.0 [7.8 to 8.3] | 8.6 [8.1 to 9.1]

4. Secondary Outcome: Number of Carbohydrate Treatments
Description: Assess the number of rescue carbohydrate treatments.
Time Frame: Entire 21 hour study duration excluding the first four hours
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: carbohydrate treatments
Arm/Group | Standard Insulin Pump Therapy | Closed-loop Without Adjustment | Closed-loop With Adjustment
Number analyzed (Participants) | 21 | 21 | 21
carbohydrate treatments | 0.33 [0.09 to 0.58] | 0.43 [0.15 to 0.71] | 0.29 [0.06 to 0.51]

5. Secondary Outcome: Percent of Time With Sensed Glucose < 50 mg/dl
Description: Assess the percent of time that the Dexcom G4 or G4 Share reported sensor glucose values less than 50 mg/dl using Dexcom sensor downloads.
Time Frame: Entire 21 hour study duration excluding the first four hours
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: percent of time
Arm/Group | Standard Insulin Pump Therapy | Closed-loop Without Adjustment | Closed-loop With Adjustment
Number analyzed (Participants) | 21 | 21 | 21
percent of time | 0.001 [0.000 to 0.03] | 0.001 [0.000 to 0.002] | 0.0 [0.000 to 0.00]

6. Secondary Outcome: Percent of Time With Sensed Glucose > 180 mg/dl
Description: Assess the percent of time that the Dexcom G4 or G4 Share reported sensor glucose values greater than 180 mg/dl using Dexcom sensor downloads.
Time Frame: Entire 21 hour study duration excluding the first four hours
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: percent of time
Arm/Group | Standard Insulin Pump Therapy | Closed-loop Without Adjustment | Closed-loop With Adjustment
Number analyzed (Participants) | 21 | 21 | 21
percent of time | 26.9 [19.8 to 34.1] | 16.9 [13.2 to 20.6] | 25.2 [18.7 to 31.7]

7. Secondary Outcome: Number of Events Capillary Blood Glucose (CBG) <70 mg/dl
Description: Number of events measured with capillary blood glucose <70 mg/dl.
Time Frame: Entire 21 hour study duration excluding the first four hours
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: occurrences of blood glucose < 70 mg/dl
Arm/Group | Standard Insulin Pump Therapy | Closed-loop Without Adjustment | Closed-loop With Adjustment
Number analyzed (Participants) | 21 | 21 | 21
occurrences of blood glucose < 70 mg/dl | 0.43 [0.15 to 0.71] | 0.33 [0.09 to 0.58] | 0.24 [0.03 to 0.45]

8. Secondary Outcome: Number of Events With CBG Between 70 - 180 mg/dl
Description: Assess the number of events that the Contour Next BG meter reported blood glucose values between 70-180 mg/dl using meter downloads.
Time Frame: Entire 21 hour study duration excluding the first four hours
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: # of events
Arm/Group | Standard Insulin Pump Therapy | Closed-loop Without Adjustment | Closed-loop With Adjustment
Number analyzed (Participants) | 21 | 21 | 21
# of events | 1.6 [1.3 to 1.9] | 3.1 [2.7 to 3.5] | 3.0 [2.6 to 3.4]

9. Secondary Outcome: Number of Events With CBG <50 mg/dl
Description: Assess the total number of events that the Contour Next BG meter reported blood glucose values less than 50 mg/dl across all participants in each group.
Time Frame: Entire 21 hour study duration excluding the first four hours
Population: as for outcome 1
Measure: Number; unit: occurrences of blood glucose < 50 mg/dl
Arm/Group | Standard Insulin Pump Therapy | Closed-loop Without Adjustment | Closed-loop With Adjustment
Number analyzed (Participants) | 21 | 21 | 21
occurrences of blood glucose < 50 mg/dl | 1 | 0 | 1

10. Secondary Outcome: Percent of Time of CBG>180 mg/dl
Description: Assess the percent of time that the Contour Next BG meter reported blood glucose values greater than 180 mg/dl using meter downloads.
Time Frame: Entire 21 hour study duration excluding the first four hours
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: percentage of time
Arm/Group | Standard Insulin Pump Therapy | Closed-loop Without Adjustment | Closed-loop With Adjustment
Number analyzed (Participants) | 21 | 21 | 21
percentage of time | 1.1 [0.7 to 1.4] | 0.7 [0.4 to 1.0] | 1.1 [0.6 to 1.6]

ADVERSE EVENTS:
Time Frame: 9 months
Arm/Group | Standard Insulin Pump Therapy | Closed-loop Without Adjustment | Closed-loop With Adjustment
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/23 | 0/23
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/23 | 0/23
Other Adverse Events (participants affected / at risk) | 1/23 | 3/23 | 3/23
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard Insulin Pump Therapy (N=23) | Closed-loop Without Adjustment (N=23) | Closed-loop With Adjustment (N=23)
nausea (Gastrointestinal disorders) | 1 (1) | 2 (2) | 2 (2)
mild edema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
headache (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
chills (General disorders) | 0 (0) | 0 (0) | 1 (1)
ligh headedness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes